CLINICAL TRIAL: NCT03301493
Title: The Use of Genomic Testing and the Resulting Medical Decisions According to Target Identification
Brief Title: Genomic Testing and Resulting Medical Decisions
Status: Completed | Type: Observational
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Roche Pharma AG (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: AGMT_NGS-Registry
Record Dates: First submitted 2017-09-22; First posted 2017-10-04 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Cancer of Unknown Origin; Cancer Refractory; Cancer of Stomach; Cancer Head Neck; Cancer of Skin; Cancer, Lung; Cancer Colorectal; Cancer of Esophagus; Cancer, Bladder; Cancer, Uterus; Cancer Cervix; Cancer Liver; Cancer, Kidney; Cancer, Breast; Hematologic Neoplasms
MeSH Terms: conditions — Neoplasms, Unknown Primary; Stomach Neoplasms; Head and Neck Neoplasms; Skin Neoplasms; Lung Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Urinary Bladder Neoplasms; Uterine Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Hepatocellular; Kidney Neoplasms; Breast Neoplasms; Hematologic Neoplasms | interventions — Genetic Profile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Genomic testing — Genomic profiling, indicated as assessed by the medical need and as deemed appropriate by the physician according to routine practice

SUMMARY:
There is no evidence available about which molecular profiling methods are currently used for cancer patients in Austrian clinical practice. The construction of the registry proposed as a completely independent research endeavor, will be helpful for scientific evaluation and the establishment of highly credible data.

DETAILED DESCRIPTION:
In the situation of enormous possible beneficial options for patients, health care systems, researchers and companies and the simultaneously present high number of uncertainties, the establishment of an independent registry for patients undergoing any type of comprehensive genomic profiling offers many advantages.

In particular, an overview of the speed of development, the "market penetration", the use of the technology in specific indications (tumor types, stages and in specific situations of unresponsiveness to certain drugs), the frequency by which treatment decisions will definitely follow the result of comprehensive genomic profiling and the reasons for this, the treatment outcome of such patients, the platform technologies applied (in-house (which types), vs. commercial) and the development of these parameters over time and in relation to the development of novel drugs will be analyzed.

The registry proposes to cover the time period from the years 2016 to 2019, which will allow for assessment of both the current and emerging landscape of genomic/molecular testing practice in Austria and effect of molecular profiling on patient care and outcome.

ELIGIBILITY:
Inclusion Criteria:

This registry will include cancer patients for which broad genomic profiling is indicated as assessed by the medical need and as deemed appropriate by the physician, for example

* cancer with high mutational load and suspicion of regular or frequent formation of neoantigens

  * skin, lung, stomach, esophagus, colorectum, bladder, uterus, cervix, liver, head and neck, kidney, breast
  * lymphoma B-cell
* any other neoplastic disease where molecular targeting is performed but treatment fails
* cancer of unknown primary origin (CUP)
* planned or already carried out comprehensive genomic testing as of Jan 1, 2016 note: this registry will not initially register patients who are tested for only 1-5 mutations by conventional means, but patients undergoing genomic profiling based on NGS)
* a patient´s signed informed consent
* Patients ≥ 18 years of age

Exclusion Criteria:

* Due to the non-interventional design of the registry there are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of oncology patients who received or plan to receive comprehensive genomic testing anytime on or after January 1, 2016. Patient medical, testing and treatment information will be obtained through extraction of data from existing patient medical charts. Longitudinal follow-up data, including survival and tumor progression, will also be extracted from patient medical charts. This patient follow-up data will be obtained until patient death or loss to follow-up.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Types of:molecular profiling methods | 3 years
  To describe types of:molecular profiling methods used in the Austrian registry centres
Types of cancer, for which comprehensive molecular profiling is used | 3 years
  To describe types of cancer, for which comprehensive molecular profiling is used
Timing of molecular profiling | 3 years
  To describe the timing of molecular profiling in relation to stage of the disease (e.g. at diagnosis, after surgery, radiation therapy, after first/second/third/late line)

SECONDARY OUTCOMES:
Number of patients with mutations identified | 3 years
  To describe targets identified:
  * number of patients with at least one mutation identified
  * number of patients with at least one druggable target identified
  * number of patients with more than one druggable targets identified
  * number of druggable targets per cancer type
Quality standards | 3 years
  To describe tests used and quality standards:
  * to compare results of NGS based molecular test systems with single marker tests or small gene panel tests
  * quality standards of the test methods used (TAT, certification status)
  * to evaluate development of methods used over time
  * usage of commercial testing vs. in-house testing, platforms used, and number of genes as well as gene size analyzed (eg whole exome with or without selected intron sequencing vs. hot spot exome sequencing)
Treatment decisions | 3 years
  To describe treatment decisions:
  * frequency by which treatment decision follows the result of NGS testing
  * frequency with druggable targets with available on-label therapy option
  * treatment decisions in the presence of more than one druggable target
Outcome of treatment | 3 years
  To describe outcome of treatment in patients receiving therapy in concordance with the test result

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, MD, Principal Investigator — IIIrd Medical Department, Private Medical University Hospital Salzburg
Locations (11):
- Austria (11):
  - IIIrd Medical Department, Private Medical University Hospital Salzburg, Salzburg, Salzburg
  - Innere Medizin II, LKH Feldkirch, Feldkirch
  - Medizinische Universitaet Graz, Univ.-Klinik f. Innere Medizin, Onkologie, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Universitätsklinikum Krems, Krems
  - BHS Linz: Interne I: Internistische Onkologie, Hämatologie und Gastroenterologie, Linz
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Medizinische Universität Wien, Vienna
  - Salzkammergut-Klinikum Vöcklabruck, Vöcklabruck
  - Klinikum Wels-Grieskirchen GmbH, Wels
  - St. Vinzenz Krankenhaus Betriebs GmbH, Zams

REFERENCES:
- [Derived] Heregger R, Huemer F, Hutarew G, Hecht S, Cheveresan L, Kotzot D, Schamschula E, Rinnerthaler G, Melchardt T, Weiss L, Greil R. Sustained response to brigatinib in a patient with refractory metastatic pheochromocytoma harboring R1192P anaplastic lymphoma kinase mutation: a case report from the Austrian Group Medical Tumor Therapy next-generation sequencing registry and discussion of the literature. ESMO Open. 2021 Aug;6(4):100233. doi: 10.1016/j.esmoop.2021.100233. Epub 2021 Aug 7. PMID 34371380